CLINICAL TRIAL: NCT00853411
Title: Th2 Effects on Eicosanoid Pathways: Implications for Altered Innate Responses in Asthma
Brief Title: Asthma Exacerbation Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by Investigator due to lack of eligible subjects.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sally E. Wenzel MD, Professor of Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO08010052
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Moderate to severe asthma
MeSH Terms: conditions — Asthma | interventions — Prednisone

INTERVENTIONS:
Drug: prednisone — Druing asthma exacerbation, subjects will be dosed to prednisone.

SUMMARY:
Asthma is a clinical syndrome that is well recognized by health care practitioners, yet asthma pathogenesis still remains poorly understood. Asthma affects approximately 20 million Americans, who suffer around 5,000 deaths annually. More than 70% of people with asthma also suffer from allergies. Although many advances in understanding the pathophysiology of asthma have been made in the past few decades, more studies are necessary to achieve a more thorough understanding of asthma at the cellular and molecular level.

The majority of murine models suggest asthma and "allergic" responses involve activation of Th2 cytokine pathways, including IL-4 and -13. Similarly in humans, several lines of evidence support a large role for Th2 adaptive immunity. These include the large majority of asthmatic patients with atopy; the measurement of increased amounts of Th2 cytokines, including IL-4 and IL-13 in the airways and sputum of mild asthma; and most recently, the observed efficacy of anti-IgE therapy in "allergic" asthma. However, other data, including the large numbers of subjects with atopy and no asthma, suggest Th2 adaptive responses are insufficient to explain many aspects of asthma. Whether and how innate and adaptive immune pathways interact in human asthma is not clear, with few studies beginning to address these interactions in vitro and in vivo.

For this reason, the investigators of this study would like to prospectively enroll patients with known asthma and follow them through an asthma exacerbation, while treating them with a standardized protocol. Over six week's duration, the investigators would like to study patients by collecting physiologic data such as spirometry, and biologic material in the form of sputum, nasal scraping, venous blood, exhaled breath and sputum. It is our aim to fully characterize the impact of the prostaglandin/cycloygenase/eicosanoid pathway as it relates to asthma exacerbation and recovery.

Completion of this study in human asthma may provide new mechanistic insights into how relationships between innate and adaptive immune responses influence the course of an asthma exacerbation. The information obtained from this research and the corresponding studies may lead to innovative medical therapies and insight into the role of the epithelium and its interactions with both innate and adaptive immunity.

ELIGIBILITY:
Inclusion Criteria:

* All adults (age 18 and older) with moderate-severe persistent asthma identified by their physicians at the Comprehensive Lung Center and UPMC network physicians, and those individuals self-referred to the asthma research center will be considered for enrollment.
* All subjects will be involved in the research design first by participating in clinical testing to characterize the absence of any respiratory disease and the severity of asthma.
* Clinical testing will include:

  * spirometry
  * methacholine challenge (when necessary for diagnosis)
  * allergy testing
  * nitric oxide monitoring.
* These tests will be performed as part of the research design on all adult subjects ages 18-60.
* Only patients on inhaled corticosteroids (CS) regularly at doses of >200 micrograms/day (fluticasone or equivalent) will be entered into the trial. There is no upper limit of CS dose.

Exclusion Criteria:

* The presence of any of the following will exclude a patient from study enrollment:

  * Subjects with mental handicaps
  * Subjects with obvious lower respiratory tract bacterial infection (pneumonia)
  * Subjects who are unable to provide consent directly and for whom an appropriate legal representative cannot be found to provide consent
  * Subjects who have previously indicated that they do not wish to be enrolled in this study.
  * A greater than five pack year history of smoking or current smoking.
  * A prior diagnosis of vocal cord dysfunction, cystic fibrosis or chronic obstructive pulmonary disorder as well as any other lung disease besides asthma, or any coronary artery disease, hypertension, diabetes or renal failure that is not well-controlled as deemed by the principal investigator.
  * Use of the 5 lipoxygenase inhibitor zileuton
  * Regular use of aspirin or other nonsteroidal anti-inflammatory (intermittent use will be allowed, but patients will be asked to take acetaminophen while in the exacerbation phase of the trial if anti-pyretic/analgesic medication is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
We will determine whether there is evidence for both adaptive and innate factors/responses in vivo at the time of an asthma exacerbation, as well as the relationship to infection.
  Our primary outcome will be differences in 15S HETE, PGE2 and their ratio in sputum of asthmatics with worsening disease (exacerbations), as compared to their stable state (resolution).